CLINICAL TRIAL: NCT00991575
Title: Long Term Vascular Changes in Type 1 Diabetes, Clinical Aspects and Biological Markers
Brief Title: Long Term Vascular Changes in Type 1 Diabetes
Acronym: DM09
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Aker (Other)
Responsible Party: Principal Investigator, Kari Anne Sveen, MD, Oslo University Hospital
Other Study IDs: 916501; S-08843c/21262
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 1; Complications; Coronary Heart Disease
Keywords: Diabetes mellitus, type1; cardiovascular disease; diabetes complications; Glycation end products, advanced
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Coronary Disease; Diabetes Mellitus; Cardiovascular Diseases; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine, tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetes, type 1

SUMMARY:
The main purpose of this study is to investigate progression of late complications of diabetes during the last ten years in a well characterized cohort of type 1 diabetes with a long duration of the disease, and to define factors responsible for the progression of late complications.

DETAILED DESCRIPTION:
Despite intensively research in the field of hyperglycaemia and coronary heart disease in type 1 diabetes it is still not known in detail how hyperglycaemia leads to damage of the vessels.

The aims of the present proposal are therefore two-fold:

1. To study in detail the progression of atherosclerosis (and micro vascular complications) in a well characterized cohort of type 1 diabetes with a long duration of the disease. This project will be a continuation of the Oslo study, a cohort started in 1982, with the last follow-up study in 1999/2000.
2. To define factors responsible for the progression of coronary heart disease (and micro vascular complications) in this cohort.

ELIGIBILITY:
The original criteria from 1982:

Inclusion Criteria:

* Age 18-45 years
* Diagnosis of type 1 diabetes at < 30 years of age, disease duration > 7 but < 30 years
* C-peptide < 0, 1 nmol/l

Exclusion Criteria:

* Serum creatinine > 150 µmol/l
* Diastolic blood pressure <100mmHg
* Overt nephropathy
* Proliferative retinopathy
* Pregnancy
* A history of neuropathy
* Other chronical disease
* Treatment with other drugs except insulin and oral contraceptives

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project will be a continuation of the previous cohort performed originally from 1982. The group or cohorts will be selected from primary care clinic.
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2009-04-01; Primary Completion 2010-05-20 (Actual); Study Completion 2010-06-20 (Actual)

PRIMARY OUTCOMES:
Fatal and non fatal cardiovascular disease (CVD) and stroke | One year

SECONDARY OUTCOMES:
Vessel area stenosis | One year

CONTACTS AND LOCATIONS:
Overall Officials: Kristian F Hanssen, Professor MD, Principal Investigator — Oslo university hospital, Aker, Norway
Locations (1):
- Oslo University hospital, Aker, Oslo, Norway